CLINICAL TRIAL: NCT06925607
Title: A Phase l Clinical Study Evaluating the Distribution and Dynamic Behavior of Nuclide Labeled TH-SC01 Cells in Vivo in Patients With Radiation Proctitis
Brief Title: Evaluate the Distribution and Dynamic Behavior of Nuclide Labeled TH-SC01 Cells in Vivo in Patients With Radiation Proctitis
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Topcel-KH Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TH-SC01-RP-Ⅰ-05
Record Dates: First submitted 2025-04-07; First posted 2025-04-13 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Radiation Proctitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- MSCs treatment group (Experimental)
  Interventions: Drug: Mesenchymal Stem Cells (MSCs)

INTERVENTIONS:
Drug: Mesenchymal Stem Cells (MSCs) — single dose injection (120 million cells)

SUMMARY:
A Phase l clinical study evaluating the distribution and dynamic behavior of Nuclide labeled TH-SC01 cells in vivo in patients with Radiation proctitis

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Good physical condition (WHO performance status score 0-1).
3. Patient received radiotherapy after being pathologically diagnosed with pelvic malignant tumors
4. Patient diagnosed with chronic radiation proctitis after undergoing colonoscopy more than 6 months after the completion of radiotherapy and did not respond to conventional treatment.
5. The LENT-SOMA score was ≥1 during the screening period.
6. All subjects and their partners were not planning to have a child from screening to the end of the trial and agreed to use effective non-drug contraception during the trial.

Exclusion Criteria:

1. Patients with severe, progressive and uncontrollable diseases of the liver, blood, gastrointestinal tract, endocrine system, lungs, heart, nervous system, mental system or brain.
2. Patients with allergic constitution or severe systemic autoimmune diseases.
3. Patients with active massive gastrointestinal bleeding or acute intestinal obstruction during the screening period.
4. Pregnant or lactating women.
5. Patients with rectal stenosis or fistula formation that restricts endoscopic treatment and require surgical treatment.
6. Patients with a LENT-SOMA score of 4 during the screening period.
7. Serum virology test (HBeAg, HCV antibody, HlV antibody, Treponema pallidum antibody) positive.
8. Patients with uncontrolled tumors, tumor recurrence or metastasis.
9. Subjects received any investigational drug within 3 months prior to the screening.
10. Subjects received stem cell treatment.
11. Participants considered inappropriate to participate in this clinical trial

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Radioactive distribution | 8-12 hour、32-36 hour、 56-60 hour. 104-108 hour、152-156 hour, 296-300 hour
  The radioactive distribution in the injection site and various organs or tissues after local injection in patients with radiation proctitis

SECONDARY OUTCOMES:
Safety endpoint: Treatment-related adverse events/adverse reactions, serious adverse events/serious adverse events | Week1, Week 4, Week 24，Month 24
  All subjects were observed for any adverse events/reactions or serious adverse events/reactions that occurred during the clinical trial, including but not limited to clinically significant abnormal changes in clinical symptoms, physical examination, vital signs examination, laboratory examination, 12- ead electrocardiogram examination, etc. The clinical features, severity, occurrence time, end time, treatment and outcome of the disease should be recorded, and the correlation between the disease and the investigational drug should be determined.
Effectiveness endpoint:Clinical symptom assessment, endoscopic evaluation and clinical improvement. | Week 4，Week 24
  The clinical symptom assessment adopts the LENT-SOMA score， total score ranges from 0 to 4, higher score means more severe symptoms.
  The endoscopic evaluation adopts the Vienna Rectoscopy Score, The score range from 0 to 5 points. The highest score of each individual item is counted as the total VRS score. Higher the VRS score means more severe lesions.
Radiation exposure | Week 1
  The uptake rate (%ID), absorbed dose and whole-body effective dose of important organs or tissues after local injection administration of [89Zr] human-derived TH-SC01 cell injection.